CLINICAL TRIAL: NCT07279012
Title: Exploring the Potential of Minimally Invasive Le Fort I Approach to Enhance Patient Outcomes
Brief Title: Minimally Invasive Le Fort I Osteotomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, İbrahim Mert Erkan, resident, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2022/190
Record Dates: First submitted 2025-12-01; First posted 2025-12-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Orthognathic Surgical Procedures
Keywords: minimally invasive; le fort I osteotomy; orthognathic surgery; patient outcomes; enhanced recovery

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Minimally Invasive Le Fort I Osteotomy (Experimental)
  Interventions: Procedure: Minimally Invasive Le Fort I Osteotomy
- Conventional Le Fort I Osteotomy (Active Comparator)
  Interventions: Procedure: Conventional Le Fort I Osteotomy

INTERVENTIONS:
Procedure: Minimally Invasive Le Fort I Osteotomy — Patients in this arm undergo the minimally invasive Le Fort I osteotomy (MI-Le Fort I). The procedure involves limited mucosal incision and soft tissue dissection. The pterygomaxillary separation is achieved through a frontal approach without osteotomizing the pterygoid plates. This technique aims to reduce surgical morbidity, intraoperative bleeding, and postoperative swelling compared to the conventional Le Fort I osteotomy.
  Arms: Minimally Invasive Le Fort I Osteotomy
Procedure: Conventional Le Fort I Osteotomy — Patients in this arm undergo the conventional Le Fort I osteotomy technique. The procedure includes standard wide mucoperiosteal flap elevation and lateral maxillary wall exposure, followed by pterygomaxillary separation using a curved osteotome and mallet. This approach serves as the control group for comparison with the minimally invasive technique.
  Arms: Conventional Le Fort I Osteotomy

SUMMARY:
This is a single-center, prospective, randomized, controlled, and double-blind clinical study designed to evaluate the clinical outcomes of the minimally invasive Le Fort I osteotomy (MI-Le Fort I) compared with the conventional Le Fort I osteotomy (Le Fort I) in patients undergoing orthognathic surgery.

Patients aged 18 to 40 years, classified as ASA I, will be randomly assigned to one of two groups: the MI-Le Fort I group or the Le Fort I group. Intraoperative parameters including blood loss (mL) and operative time (minutes) will be recorded. Postoperative facial swelling will be assessed using three-dimensional stereophotogrammetry, pain intensity will be measured with a visual analog scale (VAS). Additional outcomes will include hospitalization time, early recovery of upper lip sensation assessed by the pinprick test, and pterygomaxillary separation patterns evaluated using postoperative CBCT imaging.

The aim of this study is to compare the clinical outcomes of the MI-Le Fort I approach with the Le Fort I approach under controlled conditions. The study hypothesizes that the MI-Le Fort I osteotomy improves patient outcomes by minimizing soft tissue trauma without compromising surgical effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent Le Fort I osteotomy for maxillary dentofacial deformity
* Patients classified as ASA I
* Patients over 18 years of age

Exclusion Criteria:

* Patients with uncontrolled diabetes
* Patients with metabolic bone diseases (e.g., hyperparathyroidism, Paget's disease)
* Patients with syndromic conditions (e.g., Pierre Robin syndrome, Treacher Collins syndrome)
* Patients who had previously undergone maxillary surgery due to trauma, tumors, or cysts and had sequelae involving the upper jaw
* Patients with a history of previous orthognathic surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2022-02-24 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
Operative Time | Intraoperative period (from mucosal incision to final suture placement)
  Operative time will be measured in minutes, from the initial mucosal incision to the final suture placement, using a chronometer.
Bleeding | Intraoperative period (from mucosal incision to final suture placement)
  Bleeding volume will be measured in milliliters from the initial mucosal incision to the final suture placement, using a calibrated aspirator.
Postoperative Edema | Postoperative days 1, 7, 14, 30 and 90
  The 3dMD imaging system (3dMD, Atlanta, GA, USA) and 3dMD Vultus software were used to evaluate the amount of postoperative edema. Three-dimensional images were taken with the teeth in maximum intercuspation, lips relaxed, and eyes open on postoperative days 1, 7, 14, 30, and 90. Edema was calculated separately for the right and left sides and was recorded as surface area in square centimeters (cm²).
Postoperative Pain | Postoperative hours 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11 and 12
  Postoperative pain was evaluated using the Visual Analogue Scale for the right and left sides separately. In this scale, '0' meant no pain, and '100' represented maximum pain. Patients were questioned at postoperative 1st, 2nd, 3rd, 4th, 5th, 6th, 7th, 8th, 9th, 10th, 11th and 12th hours, and the results were recorded in the patient follow-up form.

SECONDARY OUTCOMES:
Hospitalization | From the end of surgery until hospital discharge (typically within 48 hours)
  The total postoperative hospitalization time (in hours) will be recorded for each participant. The measurement will cover the period from the end of surgery until hospital discharge.
Pterygomaxillary Separation Pattern | Postoperative first day
  The pterygomaxillary separation pattern will be evaluated using postoperative cone-beam computed tomography (CBCT) images. Each side will be classified according to the type of separation between the maxillary tuberosity and the pterygoid plates. The assessment aims to compare the frequency and characteristics of separation types between the minimally invasive Le Fort I osteotomy and the conventional Le Fort I osteotomy groups.
Neurosensory Test: Upper Lip Sensation Recovery | Postoperative days 7, 14, and 30
  Recovery of upper lip sensation will be evaluated using the pinprick test applied bilaterally in the upper lip region. Each side will be scored on a five-point ordinal scale to determine the degree of infraorbital nerve recovery.

CONTACTS AND LOCATIONS:
Locations (1):
- Erciyes University Faculty of Dentistry Department of Oral and Maxillofacial Surgery, Kayseri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No